CLINICAL TRIAL: NCT02568371
Title: Biobank Based on the i-Share Student Cohort
Acronym: bio-Share
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2015/07
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: biobank; DNA; genetic; young adults; cohort study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma ; serum ; whole blood ; red blood cells ; DNA ; RNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The bio-Share project aims at collecting blood samples in students participating in the i-Share cohort (www.i-share.fr). Investigators aim at setting up a platform that will enable investigators in the future to study biological determinants of conditions that affect young adults and to test certain hypotheses on the pathophysiology and mechanisms underlying diseases occurring both at a young age and later in life (as early exposures may also impact late onset diseases)

DETAILED DESCRIPTION:
The i-Share cohort was set up to study various important aspects of students' health and to better understand early mechanisms contributing to the occurrence of common diseases representing an important public health burden. The i-Share cohort is funded by an "investment for the future grant" from the French National Research Agency (ANR-10-COHO-05-01) with the aim to recruit 30000 students at the University of Bordeaux, and a few additional partner universities in France and abroad (www.i-share.fr).

The bio-Share study is a biological repository embedded within the i-Share study, aiming at collecting blood samples (for genetic analyses as well as measurement of other biomarkers) from a subset of 2000 i-Share participants volunteering for this ancillary project.

The goal is to set up a platform that will enable investigators in the future to study biological determinants of conditions that affect young adults and to test certain hypotheses on the pathophysiology and mechanisms underlying diseases occurring both at a young age and later in life (as early exposures may also impact late onset diseases).

The biobank will comprise the following biological materials: plasma, serum, whole blood, red blood cells, DNA, RNA. Levels of fasting glucose and lipid levels (total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides) will be returned to participants.

ELIGIBILITY:
Inclusion Criteria:

* Be an i-Share participant in Bordeaux
* Being aged 18 years or more
* Being affiliated or beneficiary of a social security
* Having filled out the first online i-Share questionnaire
* Having signed a written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women,
* Persons who cannot personally give their consent and adults under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The bio-Share study is a biological repository embedded within the i-Share study, aiming at collecting blood samples from a subset of 2000 i-Share participants volunteering for this ancillary project.
Sampling Method: Probability Sample
Enrollment: 1997 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
The acquisition date of blood samples | Day 1
The number of the aliquots for each of the stored biological samples | Day 1
The total volume of the aliquots for each of the stored biological samples | Day 1

SECONDARY OUTCOMES:
Glucose (fasting) | Day 1
Total cholesterol (fasting) | Day 1
High-density lipoprotein cholesterol (fasting) | Day 1
Low-density lipoprotein-cholesterol (fasting) | Day 1
Triglycerides (fasting) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie DEBETTE, MD, PhD, Study Director — University of Bordeaux, Inserm U897, Bordeaux University Hospital; Christophe TZOURIO, MD, PhD, Study Director — University of Bordeaux, Inserm U897, Bordeaux University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux - PELLEGRIN, Bordeaux, Aquitaine, France